CLINICAL TRIAL: NCT00600457
Title: Modified Polyurethane Film Dressing For Skin Graft Donor Sites
Status: Completed | Type: Observational
Sponsor: Klinik Bogenhausen (Other)
Responsible Party: Ulf Dornseifer, MD, Department of Plastic Surgery, Academic Hospital Munich-Bogenhausen, Technical University Munich
Other Study IDs: MOPS-1
Record Dates: First submitted 2008-01-23; First posted 2008-01-25 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Wound Healing
Keywords: healing time; pain; infection
MeSH Terms: conditions — Pain; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A,1
  Interventions: Device: Polyurethane Film

INTERVENTIONS:
Device: Polyurethane Film — The modified polyurethane film is combined with a secondary absorbent dressing and remained intact until the 10th postoperative day

SUMMARY:
The purpose of this study is to determine whether the combination of modified polyurethane film and secondary absorbent dressing for skin graft donor sites avoids the regular uncontrolled leakage, but holds up the advantages of film dressings for this kind of wound.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18 who require skin grafting

Exclusion Criteria:

* Individuals under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
uncontrolled leakage | 1-10th day postoperative

SECONDARY OUTCOMES:
pain | 1-10th day postoperative
infection | 1-10th day postoperative
epithelization status | 10th day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Dornseifer, MD, Principal Investigator — Department of Plastic, Reconstructive, Hand and Burn Surgery, Academic Hospital Munich-Bogenhausen, Technical University Munich
Locations (1):
- Department of Plastic, Reconstructive, Hand and Burn Surgery, Academic Hospital Munich Bogenhausen, Technical University Munich, Munich, Germany

REFERENCES:
- [Background] Birdsell DC, Hein KS, Lindsay RL. The theoretically ideal donor site dressing. Ann Plast Surg. 1979 Jun;2(6):535-7. doi: 10.1097/00000637-197906000-00015. PMID 396845
- [Background] James JH, Watson AC. The use of Opsite, a vapour permeable dressing, on skin graft donor sites. Br J Plast Surg. 1975 Apr;28(2):107-10. PMID 1098708
- [Background] Ramirez OM, Granick MS, Futrell JW. Optimal wound healing under Op-Site dressing. Plast Reconstr Surg. 1984 Mar;73(3):474-5. doi: 10.1097/00006534-198403000-00028. PMID 6701224
- [Background] Barnea Y, Amir A, Leshem D, Zaretski A, Weiss J, Shafir R, Gur E. Clinical comparative study of aquacel and paraffin gauze dressing for split-skin donor site treatment. Ann Plast Surg. 2004 Aug;53(2):132-6. doi: 10.1097/01.sap.0000112349.42549.b3. PMID 15269581